CLINICAL TRIAL: NCT00908804
Title: Open Versus Laparoscopic Appendectomy in Suspected Acute Appendicitis - a Prospective Randomised Clinical Trial With With 10-Year Follow-up
Brief Title: Open Versus Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Other Study IDs: NKCH-surg-004
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Appendicitis
Keywords: acute appendicitis
MeSH Terms: conditions — Appendicitis

ARMS (2):
- open appendectomy (Active Comparator)
  Interventions: Procedure: open appendectomy
- laparoscopic appendectomy (Active Comparator)
  Interventions: Procedure: laparoscopic appendectomy

INTERVENTIONS:
Procedure: open appendectomy
  Arms: open appendectomy
Procedure: laparoscopic appendectomy
  Arms: laparoscopic appendectomy

SUMMARY:
The aim of this prospective randomized trial is to compare the feasibility of open with laparoscopic appendectomy in suspected acute appendicitis. The investigators especially focused on the postoperative recovery and long-term complications.

ELIGIBILITY:
Inclusion Criteria:

* age over 15 years
* suspected acute appendicitis
* suitability for laparoscopy

Exclusion Criteria:

* patients refusal to participate
* lack of a laparoscopic surgeon

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
Complication; wound problem or other primary complication

CONTACTS AND LOCATIONS:
Locations (1):
- North Karelia Central Hospital, Clinic of Surgery, Joensuu, Finland

REFERENCES:
- [Derived] Kouhia ST, Heiskanen JT, Huttunen R, Ahtola HI, Kiviniemi VV, Hakala T. Long-term follow-up of a randomized clinical trial of open versus laparoscopic appendicectomy. Br J Surg. 2010 Sep;97(9):1395-400. doi: 10.1002/bjs.7114. PMID 20632312